CLINICAL TRIAL: NCT02969473
Title: Definitive Concurrent Chemoradiotherapy With Docetaxel Plus Cisplatin Versus 5-fluorouracil Plus Cisplatin in Patients With Esophageal Squamous Cell Carcinoma: a Phase II Randomized Controlled Trial
Brief Title: Definitive Concurrent Chemoradiotherapy With Docetaxel Plus Cisplatin Versus 5-fluorouracil Plus Cisplatin in Patients With Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhu Yujia (Other)
Responsible Party: Sponsor-Investigator, Zhu Yujia, MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YP2010138
Record Dates: First submitted 2016-11-11; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Esophageal Neoplasm; Chemoradiation
Keywords: esophageal squamous cell carcinoma; concurrent chemoradiotherapy; docetaxel; cisplatin; 5-fluorouracil
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF group (Active Comparator): This is the active comparator group. All patients in this group will receive concurrent chemoradiotherapy with PF regimen (5-fluorouracil plus cisplatin).
  Interventions: Drug: Fluorouracil
- DP group (Experimental): This is the experimental group. All patients in this group will receive concurrent chemoradiotherapy with DP regimen (docetaxel plus cisplatin).
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Radiotherapy: All patients underwent conventional radiotherapy, 1.8-2.0 Gy per fraction and 5 fractions per week. The prescribed dose was 60-64 Gy to PTV1 and 50 Gy to PTV2. Patients received either three-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated radiation therapy (IMRT). 3D-CRT treatment plans were calculated by Pinnacle planning system and IMRT treatment plans were calculated by Monacle planning system. All patients were treated with a 6-MV or 8-MV linear accelerator.
  Chemotherapy: All patients received two cycles of chemotherapy concurrently with radiotherapy. Patients assigned to the DP group received two cycles of DP regimen (docetaxel 60 mg/m2 delivered on day 1 and cisplatin 80 mg/m2 delivered on day 1) at a 3-week interval. In cases of grade 4 hematologic toxicity or severe non-hematologic toxicities, dose adjustment was performed in the subsequent chemotherapy cycle.
  Other Names: cisplatin
  Arms: DP group
Drug: Fluorouracil — Radiotherapy: All patients underwent conventional radiotherapy, 1.8-2.0 Gy per fraction and 5 fractions per week. The prescribed dose was 60-64 Gy to PTV1 and 50 Gy to PTV2. Patients received either three-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated radiation therapy (IMRT). 3D-CRT treatment plans were calculated by Pinnacle planning system and IMRT treatment plans were calculated by Monacle planning system. All patients were treated with a 6-MV or 8-MV linear accelerator.
  Chemotherapy: All patients received two cycles of chemotherapy concurrently with radiotherapy. Patients assigned to the PF group received two cycles of PF regimen (cisplatin 80 mg/m2 delivered on day 1 and 5-FU 1000 mg/m2 continuous infusion over 24 hours daily on days 1-4) at a 3-week interval. In cases of grade 4 hematologic toxicity or severe non-hematologic toxicities, dose adjustment was performed in the subsequent chemotherapy cycle.
  Other Names: cisplatin
  Arms: PF group

SUMMARY:
In this phase II study, the investigators aim to evaluated the efficacy and toxicity of definitive concurrent chemoradiotherapy (CCRT) with docetaxel plus cisplatin (DP regimen) versus 5-fluorouracil plus cisplatin (PF regimen) in patients with esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
Esophageal cancer is one of the most fatal malignancies worldwide. Radical surgery has been the primary treatment for patients with resectable esophageal cancer. For medically unfit patients or medically fit patients who decline surgery, definitive radiotherapy plus concurrent chemotherapy has been established as a standard treatment. Since the 1980' s, the most widely used chemotherapeutic regimen in combination with radiotherapy for esophageal cancer was cisplatin (CDDP) plus 5-fluorouracil (5-FU) (the PF regimen). However, locoregionally persistent or recurrent diseases were still quite common and survival remained poor. Several previous studies conducted by the radiation therapy oncology group (RTOG) explored the efficacy of radiation dose escalation, but all results turned out disappointing. And studies incorporating intensified PF regimen or new-generation cytotoxic agents such as paclitaxel and oxaliplatin did not show any advantage over the standard-dosage PF regimen either. In this phase II study, the investigators aim to evaluated the efficacy and toxicity of definitive concurrent chemoradiotherapy (CCRT) with docetaxel plus cisplatin (DP regimen) versus 5-fluorouracil plus cisplatin (PF regimen) in patients with esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically proven squamous cell carcinoma of the esophagus
* stage II-IVA disease, including metastatic celiac or cervical nodes, according to the sixth edition of American Joint Committee on Cancer (AJCC) staging system for esophageal cancer
* aged between 18 and 70 years
* Karnofsky Performance Status (KPS) score ≥ 70
* adequate bone marrow function (leukocyte count ≥ 4000/uL, platelet count ≥ 100,000/uL), adequate liver function (serum alanine aminotransferase (ALT) level and serum aspartate aminotransferase (AST) level < twice the upper limit of normal, and serum bilirubin level of <1.5 mg/dL), and adequate renal function (creatinine clearance ≥ 50 mL/min)
* no other serious medical conditions
* life expectancy ≥ 3 months
* written informed consent

Exclusion Criteria:

* detection of distant metastasis (excluding metastatic celiac or cervical nodes) before treatment before treatment
* known allergy to CDDP, 5-FU, or docetaxel
* pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-10; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the date of randomization until the date of death, up to 5 years.

SECONDARY OUTCOMES:
Treatment response rate | From the date of randomization until six weeks after treatment completion.
Progress Free Survival (PFS) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
Acute treatment-related toxicities | From the date of randomization until six months after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghong Hu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- SYSU Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ruppert BN, Watkins JM, Shirai K, Wahlquist AE, Garrett-Mayer E, Aguero EG, Sherman CA, Reed CE, Sharma AK. Cisplatin/Irinotecan versus carboplatin/paclitaxel as definitive chemoradiotherapy for locoregionally advanced esophageal cancer. Am J Clin Oncol. 2010 Aug;33(4):346-52. doi: 10.1097/COC.0b013e3181aaca26. PMID 19841574
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Herskovic A, Martz K, al-Sarraf M, Leichman L, Brindle J, Vaitkevicius V, Cooper J, Byhardt R, Davis L, Emami B. Combined chemotherapy and radiotherapy compared with radiotherapy alone in patients with cancer of the esophagus. N Engl J Med. 1992 Jun 11;326(24):1593-8. doi: 10.1056/NEJM199206113262403. PMID 1584260
- [Background] al-Sarraf M, Martz K, Herskovic A, Leichman L, Brindle JS, Vaitkevicius VK, Cooper J, Byhardt R, Davis L, Emami B. Progress report of combined chemoradiotherapy versus radiotherapy alone in patients with esophageal cancer: an intergroup study. J Clin Oncol. 1997 Jan;15(1):277-84. doi: 10.1200/JCO.1997.15.1.277. PMID 8996153
- [Background] Gaspar LE, Winter K, Kocha WI, Coia LR, Herskovic A, Graham M. A phase I/II study of external beam radiation, brachytherapy, and concurrent chemotherapy for patients with localized carcinoma of the esophagus (Radiation Therapy Oncology Group Study 9207): final report. Cancer. 2000 Mar 1;88(5):988-95. PMID 10699886
- [Background] Minsky BD, Neuberg D, Kelsen DP, Pisansky TM, Ginsberg R, Benson A 3rd. Neoadjuvant chemotherapy plus concurrent chemotherapy and high-dose radiation for squamous cell carcinoma of the esophagus: a preliminary analysis of the phase II intergroup trial 0122. J Clin Oncol. 1996 Jan;14(1):149-55. doi: 10.1200/JCO.1996.14.1.149. PMID 8558190
- [Background] Ajani JA, Winter K, Komaki R, Kelsen DP, Minsky BD, Liao Z, Bradley J, Fromm M, Hornback D, Willett CG. Phase II randomized trial of two nonoperative regimens of induction chemotherapy followed by chemoradiation in patients with localized carcinoma of the esophagus: RTOG 0113. J Clin Oncol. 2008 Oct 1;26(28):4551-6. doi: 10.1200/JCO.2008.16.6918. Epub 2008 Jun 23. PMID 18574157
- [Background] Mason KA, Hunter NR, Milas M, Abbruzzese JL, Milas L. Docetaxel enhances tumor radioresponse in vivo. Clin Cancer Res. 1997 Dec;3(12 Pt 1):2431-8. PMID 9815644
- [Background] Hennequin C, Giocanti N, Favaudon V. Interaction of ionizing radiation with paclitaxel (Taxol) and docetaxel (Taxotere) in HeLa and SQ20B cells. Cancer Res. 1996 Apr 15;56(8):1842-50. PMID 8620502
- [Background] Li QQ, Liu MZ, Hu YH, Liu H, He ZY, Lin HX. Definitive concomitant chemoradiotherapy with docetaxel and cisplatin in squamous esophageal carcinoma. Dis Esophagus. 2010 Apr;23(3):253-9. doi: 10.1111/j.1442-2050.2009.01003.x. Epub 2009 Aug 28. PMID 19732130
- [Background] Einzig AI, Neuberg D, Remick SC, Karp DD, O'Dwyer PJ, Stewart JA, Benson AB 3rd. Phase II trial of docetaxel (Taxotere) in patients with adenocarcinoma of the upper gastrointestinal tract previously untreated with cytotoxic chemotherapy: the Eastern Cooperative Oncology Group (ECOG) results of protocol E1293. Med Oncol. 1996 Jun;13(2):87-93. doi: 10.1007/BF02993858. PMID 9013471
- [Background] Ohtsu A, Boku N, Muro K, Chin K, Muto M, Yoshida S, Satake M, Ishikura S, Ogino T, Miyata Y, Seki S, Kaneko K, Nakamura A. Definitive chemoradiotherapy for T4 and/or M1 lymph node squamous cell carcinoma of the esophagus. J Clin Oncol. 1999 Sep;17(9):2915-21. doi: 10.1200/JCO.1999.17.9.2915. PMID 10561371
- [Background] Minsky BD, Neuberg D, Kelsen DP, Pisansky TM, Ginsberg RJ, Pajak T, Salter M, Benson AB 3rd. Final report of Intergroup Trial 0122 (ECOG PE-289, RTOG 90-12): Phase II trial of neoadjuvant chemotherapy plus concurrent chemotherapy and high-dose radiation for squamous cell carcinoma of the esophagus. Int J Radiat Oncol Biol Phys. 1999 Feb 1;43(3):517-23. doi: 10.1016/s0360-3016(98)00463-5. PMID 10078631
- [Background] Chandra A, Guerrero TM, Liu HH, Tucker SL, Liao Z, Wang X, Murshed H, Bonnen MD, Garg AK, Stevens CW, Chang JY, Jeter MD, Mohan R, Cox JD, Komaki R. Feasibility of using intensity-modulated radiotherapy to improve lung sparing in treatment planning for distal esophageal cancer. Radiother Oncol. 2005 Dec;77(3):247-53. doi: 10.1016/j.radonc.2005.10.017. Epub 2005 Nov 17. PMID 16298001
- [Background] Wu VW, Kwong DL, Sham JS. Target dose conformity in 3-dimensional conformal radiotherapy and intensity modulated radiotherapy. Radiother Oncol. 2004 May;71(2):201-6. doi: 10.1016/j.radonc.2004.03.004. PMID 15110454
- [Background] Wu Q, Manning M, Schmidt-Ullrich R, Mohan R. The potential for sparing of parotids and escalation of biologically effective dose with intensity-modulated radiation treatments of head and neck cancers: a treatment design study. Int J Radiat Oncol Biol Phys. 2000 Jan 1;46(1):195-205. doi: 10.1016/s0360-3016(99)00304-1. PMID 10656393
- [Background] Katsumata N, Yasuda M, Takahashi F, Isonishi S, Jobo T, Aoki D, Tsuda H, Sugiyama T, Kodama S, Kimura E, Ochiai K, Noda K; Japanese Gynecologic Oncology Group. Dose-dense paclitaxel once a week in combination with carboplatin every 3 weeks for advanced ovarian cancer: a phase 3, open-label, randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1331-8. doi: 10.1016/S0140-6736(09)61157-0. Epub 2009 Sep 18. PMID 19767092
- [Derived] Jiang H, Makelike K, Chen B, Xi M, Li Q, Hu Y, Zhu Y. Definitive concurrent chemoradiotherapy with docetaxel plus cisplatin versus 5-fluorouracil plus cisplatin in patients with esophageal squamous cell carcinoma: long-term follow-up results of a phase II randomized controlled trial. Radiat Oncol. 2023 Sep 12;18(1):150. doi: 10.1186/s13014-023-02339-9. PMID 37700348